CLINICAL TRIAL: NCT02143531
Title: Intravenous Haloperidol Versus Ondansetron for Treatment of Established Nausea and Vomiting in Patients Undergoing Surgery With General Anesthesia: A Randomized Clinical Trial
Brief Title: Intravenous Haloperidol Versus Ondansetron for Treatment of Established Post-operative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Marie Awad, Professor of Clinical Specialty, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANES.MA 09
Record Dates: First submitted 2014-05-15; First posted 2014-05-21 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Active Comparator): Patients will receive 4 mg of Ondansetron IV upon occurrence of nausea or vomiting
  Interventions: Drug: 4 mg of Ondansetron IV
- Group II (Active Comparator): Patients will receive 1mg of Haloperidol IV upon occurrence of nausea or vomiting
  Interventions: Drug: 1mg of Haloperidol IV

INTERVENTIONS:
Drug: 4 mg of Ondansetron IV
  Arms: Group I
Drug: 1mg of Haloperidol IV
  Arms: Group II

SUMMARY:
This study aims to prove that at a dose of 1 mg Haloperidol possesses a high success rate in controlling established postoperative nausea and vomiting (PONV) in the first 24 hours following administration similar to the standard of care ondansetron 4 mg.

DETAILED DESCRIPTION:
Patients undergoing surgery under general anesthesia may experience several complications in their postoperative period. Nausea and vomiting are some of the more common of these complications. Several medications can be used for prevention of these specific complications, but treatment remains more cost-efficient.

Haloperidol is anti-psychotic which, at low doses, can prevent the occurrence of nausea and vomiting. Its usefulness for prophylaxis has been demonstrated in several studies. However, its use for treating established postoperative nausea and vomiting (PONV) has not been properly studied.

In a prospective randomized clinical trial involving adult patients undergoing elective surgery under general anesthesia, investigators will enroll 120 patients, and compare the effect of a dose of 1 mg Haloperidol versus Ondansetron 4 mg and document the varying degrees of success in treating nausea and vomiting as well as possible side effects.

Investigators expect to observe that Haloperidol is as effective as treatment with Ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80
* ASA class I, II, and III
* undergoing elective surgery under general anesthesia

Exclusion Criteria:

* Patients with history of arrhythmias, QTc prolongation or allergies to the study drugs will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The success of the anti-emetic administered in treating the postoperative nausea and vomiting (PONV) | during the first hour postoperatively
  Investigators will assess the success rate of the anti-emetic used: resolution of post-operative nausea and vomiting within 30 minutes from the adminstration of the anti-emetic will be considered "success".

SECONDARY OUTCOMES:
Severity of postoperative nausea and vomiting (PONV) | during the first 24 hours postoperatively
  Investigators will ask patients to grade the severity of their nausea episodes using the following scale:
  0. No nausea; 1. mild ; 2. Discomforting; 3. Distressing; 4. Horrible; 5. Worst possible
Recurrence of postoperative nausea and vomiting (PONV) | during first 24 hours postoperatively
Side effects in PACU | 1 hour postoperatively
  Headache, Dizzines / Vertigo, Restlessness, Nystagmus or other extra-pyramidal symptoms, Sedation highest score, Pain highest score, QT prolongation
Patient satisfaction | 24 hours after surgery
  24 hours following surgery, investigators will ask patients to grade their satisfaction with the treatment of post-operative nausea and vomiting using the following scale:
  1. Excellent; 2. Good; 3. Fair; 4. Bad
Rescue anti-emetic | during the first 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marie Aouad, MD, Principal Investigator — American Univesity of Beirut Medical Center
Locations (1):
- Marie Aouad, Beirut, Lebanon